CLINICAL TRIAL: NCT03893617
Title: Brief Stresses and DNA Integrity: An Experimental Analysis
Brief Title: Brief Stresses Experimental Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to challenges associated with the Covid-19 pandemic, we were unable to complete recruitment as planned during the period we had funding to do so.
Sponsor: Dana Bovbjerg (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Dana Bovbjerg, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO16080092; R01CA211371 (NIH)
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: DNA Damage; Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol group (Active Comparator): This group will receive a single oral dose (80mg) of propranolol in a blinded capsule during their acute stress study visit.
  Interventions: Drug: Propranolol; Behavioral: Acute stress task; Behavioral: No stress task
- Placebo group (Placebo Comparator): This group will receive a single blinded capsule containing no active medication during their acute stress study visit.
  Interventions: Drug: Placebo oral capsule; Behavioral: Acute stress task; Behavioral: No stress task

INTERVENTIONS:
Drug: Propranolol — A single oral dose (80mg) of propranolol will be administered in a blinded capsule at the start of the baseline monitoring period of the acute stress study visit.
  Arms: Propranolol group
Drug: Placebo oral capsule — A single blinded capsule containing no active medication will be administered at the start of the baseline monitoring period of the acute stress study visit.
  Arms: Placebo group
Behavioral: Acute stress task — Participants will complete speech and arithmetic tasks, performed in front of an audience (e.g., researcher staff members) and recorded by a video camera to assess non-verbal behaviors and evaluate performance. The task will be initiated following completion of baseline sample collection during the acute stress study visit and will take approximately 15 minutes.
Behavioral: No stress task — Participants will sit quietly for 5 minutes, read a short passage aloud for 5 minutes, and read a list of numbers aloud for 5 minutes. The task will be initiated following completion of baseline sample collection during the no stress study visit and will take approximately 15 minutes.

SUMMARY:
The goal of this study is to examine the impact of psychological stress on DNA integrity by conducting an experiment under controlled conditions with healthy volunteers to directly test the extent to which acute stress increases DNA damage, while simultaneously testing the blocking effects of pre-treatment with propranolol, and exploring key hypothesized mediators and moderators of the severity of the DNA damage.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-59
* Weigh at least 110 pounds
* Fasting blood sugar below 150 mg/dL, or random blood sugar below 200 mg/dL
* Thyroid stimulating hormone level between 0.25 mU/L and 6.0 mU/L
* Resting blood pressure below 160/100 mm Hg
* If female, have either regular menstrual periods (21-35 days) or are post-menopausal

Exclusion Criteria:

* Use of illicit drugs or nicotine-containing products other than cigarettes in the past month
* Current alcohol abuse
* Diagnosed with any of the following: cancer (other than basal cell skin cancer), chronic obstructive pulmonary disorder (COPD), multiple sclerosis (MS), severe traumatic brain injury, hypertension (high blood pressure), coronary artery disease, congestive heart failure, or other serious heart disease
* Current diabetes, asthma, depression, bipolar disorder, anxiety, or schizophrenia
* If female, pregnancy or breastfeeding within the past 3 months
* If female, taking any medications that prevent monthly menstrual cycles (e.g., birth control shot, IUD, "seasonal" birth control)
* Resting systolic blood pressure of < 90 mm Hg or resting pulse < 50 beats per minute

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
DNA Stress Response | Blood samples will be collected after a 60 minute baseline period and after the approximately 15 minute acute stress task period
  Change in percent tail intensity will be measured using the Comet assay of DNA damage in blood samples

SECONDARY OUTCOMES:
DNA Stress Response (8-OHdG) | Blood samples will be collected after a 60 minute baseline period and after the approximately 15 minute task period
  Change in DNA 8-OHdG levels will be measured in blood samples
DNA Stress Response (γ-H2AX) | Blood samples will be collected after a 60 minute baseline period and after the approximately 15 minute task period
  Change in cellular γ-H2AX levels will be measured in blood samples
Neuroendocrine Stress Response (Norepinephrine (NE)) | Blood samples will be collected after a 60 minute baseline period and during/after the approximately 15 minute task period
  Change in circulating plasma NE levels will be measured in blood samples
Neuroendocrine Stress Response (Epinephrine (EPI)) | Blood samples will be collected after a 60 minute baseline period and during/after the approximately 15 minute task period
  Change in circulating plasma EPI levels will be measured in blood samples
Hematological Stress Response | Blood samples will be collected after a 60 minute baseline period and after the approximately 15 minute task period
  Change in the white blood cell populations present in blood samples will be measured through complete blood count with differential analysis and flow cytometry
Cardiovascular Stress Response (Heart rate (HR)) | HR will be assessed throughout the 60 minute baseline period and during/after the approximately 15 minute task period
  Change in HR will be calculated from repeated assessments
Cardiovascular Stress Response (Systolic blood pressure (SBP)) | Blood pressure will be assessed throughout the 60 minute baseline period and during/after the approximately 15 minute task period
  Change in SBP/DBP will be calculated from repeated assessments
Cardiovascular Stress Response (Diastolic blood pressure (DBP)) | Blood pressure will be assessed throughout the 60 minute baseline period and during/after the approximately 15 minute task period
  Change in DBP will be calculated from repeated assessments
Psychological Stress Response (Anxiety Visual Analogue Scale (VAS)) | Anxiety VAS will be administered after a 60 minute baseline period and during/after completion of the tasks
  Change in anxiety levels will be assessed by self-report measure (VAS) on a 0 to 100 scale, where 0 indicates not feeling anxious and 100 indicates feeling highly anxious
Psychological Stress Response (Stress Visual Analogue Scale (VAS)) | Stress VAS will be administered after a 60 minute baseline period and during/after completion of the tasks
  Change in stress levels will be assessed by self-report measure (VAS) on a 0 to 100 scale, where 0 indicates not feeling stressed and 100 indicates feeling highly stressed

CONTACTS AND LOCATIONS:
Overall Officials: Dana Bovbjerg, PhD, Principal Investigator — University of Pittsburgh; Frank Jenkins, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States